CLINICAL TRIAL: NCT05221476
Title: RDW and CCI in the Frail Polytraumatized Patients. A Retrospective Cohort Study in a Level 1 Trauma Center.
Brief Title: Red Blood Cell Distribution Width and Charlson Comorbidity Indeces in the Frail Polytraumatized Patient.
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Valerie Weihs, MD, Medical University of Vienna
Other Study IDs: RDW Polytrauma
Record Dates: First submitted 2022-01-08; First posted 2022-02-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Polytrauma; Red Blood Cell Distribution Width; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Multiple Trauma | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- polytraumatized patients: Patients with an ISS >16 points, an AIS >3 in one body region and at least 2 different body regions affected were included.
  Interventions: Other: retrospective

INTERVENTIONS:
Other: retrospective — The investigators retrospectively analyzed the short- and long-term outcome in polytraumatized patients and the possible influence of RDW values on admission as well as preexisting comorbidities on these outcomes.

SUMMARY:
In this study patients who were admitted to our hospital with critical injuries were enrolled retrospectively from January 2012 to December 2015. Patients with an ISS>16 points, an AIS >3 in one body region and at least 2 different body regions affected were included. RDW values on admission as well as preexisting comorbidities were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ISS >16 points
* AIS >3 in one body region
* at least 2 body regions affected

Exclusion Criteria:

* patients younger than 18 years of age
* isolated traumatic brain injury
* minor injuries (AIS <3 or ISS <16 points)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of polytraumatized patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality in polytraumatized patients | January 2012 to December 2015

SECONDARY OUTCOMES:
Possible influence of RDW values (%) on admission on the long-term outcome | January 2012 to December 2015
  The influence of RDW Values (%) in polytraumatized patients on admission on the long-term outcome (late-phase death (days)) will be examined.

IPD SHARING:
Plan to Share IPD: No